CLINICAL TRIAL: NCT03832881
Title: The United Kingdom Thrombotic Thrombocytopenic Purpura Registry
Brief Title: The United Kingdom Thrombotic Thrombocytopenic Purpura Registry (UK TTP Registry)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 08/0264
Record Dates: First submitted 2019-01-11; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: TTP - Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — On Admission/Pre-treatment:
  • A 5ml double spun citrate sample (platelet free plasma separated) taken on admission and/or pre-treatment. (Part of Standard Care).
  In Remission/Approximately 3 months post admission:
  * A 5ml double spun remission citrate sample (platelet free plasma separated) following discharge from the acute episode. (Part of Standard Care)
  * A 5ml EDTA whole blood sample for DNA extraction. (Informed Consent from patient required).
  * A 5ml serum sample. (Sample taken as part of Standard Care; Informed Consent required for storage and use of sample for current and future analysis of parameters related to TTP; Current tests include, IgG subtyping and Rituximab levels.)
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: ADAMTS13, VWF assay

SUMMARY:
This is a UK (United Kingdom) based registry, involving all sites treating newly presenting Thrombotic Thrombocytopenic Purpura (TTP). From this registry, important epidemiological data will be obtained. Admission and remission samples will be collected. DNA will be collected and analysed from patients wishing to participate to determine if any link exists between mutations/polymorphisms and the risk of TTP. As part of NHS commissioning, we will be undertaking long term follow up, to understand the impact of acute TTP on morbidity and mortality.

DETAILED DESCRIPTION:
The UK TTP registry started in January 2009, following 3 years MRC funding, involving UK collaboration from all sites treating TTP patients. It has resulted in a cohort of data and samples from UK TTP cases. The registry promotes a collaborative approach with all UK patients and physicians involved with this life threatening disorder. The UK TTP registry has been used to provide information for highly specialist commissioning via NHS England and moving forward will be required to provide data relevant to the UK TTP Group and commissioners.

University College London (UCL) Haemostasis Research Unit (HRU) will collect and collate the data and help administrate for those sites participating in the registry. However, ADAMTS13 assays will no longer be subsidised. For those sites undertaking local assays, a record of cases will be shared centrally. The UK TTP registry will be part of the UK TTP Group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of TTP, defined by thrombocytopenia, MAHA which may be associated with clinical evidence of organ compromise.Confirmed by severely reduced ADAMTS13 levels and/or a positive antibody screen.
* No age restriction.
* Consent for addition to the Registry and collection/storage of admission information once in remission.
* Consent to collect, analyse and store EDTA sample once in remission.
* Consent to store samples once in remission (sample taken as part of standard care).
* For sites undertaking ADAMTS13 analysis, consent to send admission and remission samples for analysis relating to TTP.
* Follow up laboratory and clinical data at least yearly to identify any changes.

Exclusion Criteria:

* Patients with cancer or transplant associated MAHA will not be included.
* Patients not wishing to be involved with the registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting with an acute episode of Thrombotic Thrombocytopenic Purpura (TTP) will be asked to consent for the registry once in remission. However, for those sites undertaking ADAMTS13 analysis, consent for admission and remission samples for TTP cases will be requested. A screening log of all cases analysed will be kept by sites and forwarded at 3 monthly intervals. This will help identify other non-TTP causes for ADAMTS13 analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
TTP incidence | At study completion, approximately in 2023
  Number of TTP cases in the UK each year

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom